CLINICAL TRIAL: NCT05490576
Title: Pilot Phase 1 Clinical Trial of PET Scanning in Tau Protein Deposition and Connectome Analysis in Traumatic Encephalopathy Syndrome (TES) Cohort With a Probable Chronic Traumatic Encephalopathy (CTE) Pattern of Neurodegenerative Disease
Brief Title: Tau And Connectomics In TES Study
Acronym: TACIT
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Macquarie University, Australia (Other)
Collaborators: Omniscient Neurotechnology (Industry); Life Molecular Imaging GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CNTES01
Record Dates: First submitted 2022-08-04; First posted 2022-08-05 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Chronic Traumatic Encephalopathy; Traumatic Encephalopathy; Head Injury Trauma; Cognitive Impairment; Neurodegenerative Diseases
MeSH Terms: conditions — Chronic Traumatic Encephalopathy; Brain Injuries, Traumatic; Cognitive Dysfunction; Neurodegenerative Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [18F] PI-2620 PET Tau Ligand Active Agent (Experimental): Participants receive dose of active agent [18F] PI-2620 PET Tau Ligand during dynamic PET scan acquisition
  Interventions: Radiation: [18F] PI-2620 Tau Ligand

INTERVENTIONS:
Radiation: [18F] PI-2620 Tau Ligand — Tau binding ligand

SUMMARY:
This pilot study aims to assess if participants that meet the criteria for a TES diagnosis have a specific tau deposition profile on PET scanning using the PET tau binding ligand - [18F] PI-2620. It is hoped this study will highlight potential diagnostic tests of TES diagnosis, the in-life correlate of CTE.

ELIGIBILITY:
Inclusion Criteria:

* The participant must have full capacity to understand the purpose and risks of the study to provide informed consent.
* All participants must be between 40 to 70 years of age.
* Must meet the Traumatic Encephalopathy Syndrome criteria as defined by the National Institute of Neurological Disorders and Stroke Consensus Diagnostic Criteria for Traumatic Encephalopathy Syndrome, Katz. D, et. al. Neurology, 2021.
* Participants must demonstrate that they have a cognitive decline, evident by performance on neuropsychological testing.
* Standard of care blood screening within 12 months of consent to the study to exclude other medical conditions which may cause cognitive decline, such as heavy metal toxicology.
* A PET scan within 6 months of consent to the study that is not consistent with Alzheimer's disease.
* Participants must consent to undertake Positron Emission Tomography (PET) with intravenous [18F] PI-2620 PET tracer ligand.
* Participants must be able to lie still, on their back for up to 60 minutes for the scans.
* Participants must not have any metal in their bodies e.g. pacemakers, aneurysm clips which are contraindications of MRI.
* Participants must consent to the use of their medical records and medical history, including but not limited to pathology results, previous imaging results and neuropsychology results

Exclusion Criteria:

* Participants will be excluded if they do not meet all the inclusion criteria.
* Participants must not be diagnosed with or suspected to be suffering from any other neurodegenerative disease, or cerebral disease affecting cognition as identified by results of neuropsychological evaluation or neurologist consultation.
* Participants will be excluded if Staff at Macquarie Medical Imaging determine that the participant is not suitable for imaging, for any reason.
* Participants will be excluded if they have kidney and/or liver dysfunction as diagnosed by a doctor

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-02-03 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection of Tau protein 3R and 4R isoforms in patients who meet the Traumatic Encephalopathy Syndrome (TES) criteria, as defined by the National Institute of Neurological Disorders and Stroke. | 2 weeks
  Participants are either Tau positive or Tau negative, determined by the PET scan

SECONDARY OUTCOMES:
Detect disease anomalies on MRI which correlated with brain region tau deposition | 2 weeks
  Regional Tau load on PET scan compared with MRI
Compare PET tau imaging PI-2620 results in TES to prior studies in Alzheimer's disease using the same ligand | 2 weeks
  By comparing PET data against reference ranges

CONTACTS AND LOCATIONS:
Overall Officials: Rowena Mobbs, MBBS, PhD, Principal Investigator — MQ Health
Locations (1):
- Macquarie Medical Imaging, Macquarie Park, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Undecided